CLINICAL TRIAL: NCT05713578
Title: Efficacy and Safety of Apantamide Combined With Docetaxel and ADT vs. Apantamide Combined With ADT in Patients With High Tumor Burden mHSPC: a Multicenter and Prospective Cohort Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bks01
Record Dates: First submitted 2023-01-02; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Cohort Studies
Keywords: cohort study; apantamide; docetaxel; ADT

STUDY DESIGN:
Intervention Model Description: Experimental: apantamide+docetaxel+ADT;Active.Comparator: apantamide+ADT treatment
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apantamide+docetaxel+ADT (Experimental): The dosage is adjusted according to the adverse reaction (according to the instructions).Apantamide, 240 mg (4 × 60 mg tablets), once a day, orally;ADT regimen was treated with gonadotropin releasing hormone analog (GnRHa), including GnRHa agonist or GnRHa antagonist. The type, frequency and dose of ADT to be used in each research center are determined by the investigator;The treatment of docetaxel was started within 6 weeks after the treatment of apantamide and ADT. The single dose of docetaxel was 75 mg/m2, intravenous drip for 1 hour, repeated every 3 weeks, and docetaxel lasted for 6 cycles. It is up to the researcher to decide whether to use prednisone or prednisolone.
  Interventions: Drug: apantamide+docetaxel+ADT
- apantamide+ADT treatment (Active Comparator): Patients were treated with apantamide and ADT after enrollment. The patient received each drug treatment according to the instructions. The dosage is adjusted according to the adverse reaction (according to the instructions)Apantamide, 240 mg (4 × 60 mg tablets), once a day, orally;ADT regimen was treated with gonadotropin releasing hormone analog (GnRHa), including GnRHa agonist or GnRHa antagonist. The type, frequency and dose of ADT used in each research center are determined by the investigator.
  Interventions: Drug: apantamide+ADT treatment

INTERVENTIONS:
Drug: apantamide+docetaxel+ADT — Apantamide, 240 mg (4 × 60 mg tablets), once a day, orally; ADT regimen was treated with gonadotropin releasing hormone analog (GnRHa), including GnRHa agonist or GnRHa antagonist. The type, frequency and dose of ADT to be used in each research center are determined by the investigator; The treatment of docetaxel was started within 6 weeks after the treatment of apantamide and ADT. The single dose of docetaxel was 75 mg/m2, intravenous drip for 1 hour, repeated every 3 weeks, and docetaxel lasted for 6 cycles.
  Arms: apantamide+docetaxel+ADT
Drug: apantamide+ADT treatment — apantamide+ADT treatment
  Arms: apantamide+ADT treatment

SUMMARY:
This is a multicenter, prospective, cohort study to evaluate the efficacy and safety of apantamide+docetaxel+ADT versus apantamide+ADT in the treatment of patients with high tumor mHSPC.220 patients with high tumor mHSPC will be included and divided into two treatment groups according to the treatment plan:Treatment group 1: apantamide+docetaxel+ADT,Treatment group 2: apantamide+ADT treatment.The study continued treatment until the patient could not obtain clinical benefits or had intolerable toxic reactions or the patient withdrew the informed consent, whichever occurred first.

DETAILED DESCRIPTION:
This is a multicenter, prospective, cohort study to evaluate the efficacy and safety of apantamide+docetaxel+ADT versus apantamide+ADT in the treatment of patients with high tumor mHSPC.220 patients with high tumor mHSPC will be included and divided into two treatment groups according to the treatment plan:

Treatment group 1: apantamide+docetaxel+ADT

Patients were treated with apantamide+docetaxel+ADT after enrollment. The patient received each drug treatment according to the instructions. The dosage is adjusted according to the adverse reaction (according to the instructions).Apantamide, 240 mg (4 × 60 mg tablets), once a day, orally;ADT regimen was treated with gonadotropin releasing hormone analog (GnRHa), including GnRHa agonist or GnRHa antagonist. The type, frequency and dose of ADT to be used in each research center are determined by the investigator;The treatment of docetaxel was started within 6 weeks after the treatment of apantamide and ADT. The single dose of docetaxel was 75 mg/m2, intravenous drip for 1 hour, repeated every 3 weeks, and docetaxel lasted for 6 cycles. It is up to the researcher to decide whether to use prednisone or prednisolone. To prevent docetaxel related hypersensitivity and fluid retention, oral administration of 8 mg dexamethasone is recommended 12 hours, 3 hours and 1 hour before infusion of docetaxel.The study continued treatment until the patient could not obtain clinical benefits or had intolerable toxic reactions or the patient withdrew the informed consent, whichever occurred first.

Treatment group 2: apantamide+ADT treatment

Patients were treated with apantamide and ADT after enrollment. The patient received each drug treatment according to the instructions. The dosage is adjusted according to the adverse reaction (according to the instructions)Apantamide, 240 mg (4 × 60 mg tablets), once a day, orally;ADT regimen was treated with gonadotropin releasing hormone analog (GnRHa), including GnRHa agonist or GnRHa antagonist. The type, frequency and dose of ADT used in each research center are determined by the investigator.The study continued treatment until the patient could not obtain clinical benefits or had intolerable toxic reactions or the patient withdrew the informed consent, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male;
2. It was diagnosed as prostate adenocarcinoma by histological or cytological examination, and its pathological type was adenocarcinoma;
3. Bone imaging, CT or MRI showed ≥ 4 bone metastases (≥ 1 bone metastasis located outside the pelvis or spine) or visceral metastasis;
4. .Patients with recurrence after new or local treatment are sensitive to endocrine therapy;
5. Patients receiving ADT treatment (drug or surgical castration), with or without the first generation of antiandrogen drugs, for no more than 3 months, and without evidence of soft tissue imaging disease progression (according to RECIST 1.1 standard) or clinically significant PSA increase (after serum testosterone reaches the castration level, PSA increases by 50% from the lowest level), are allowed to be included in the group;
6. Plan to receive docetaxel combined with apantamide and ADT or apantamide combined with ADT;
7. ECOG PS score 0-1;
8. Adequate hematology and organ function:

   Adequate bone marrow function (no blood transfusion, no use of granulocyte colony stimulating factor): absolute neutrophil count (ANC) ≥ 1.5 × 109/L（1500/ μ L）； Hemoglobin ≥ 90 g/L (9.0 g/dL); Platelet count ≥ 100 × 109/L（100, 000/ μ L）；

   Adequate liver function: total bilirubin (TBIL) ≤ 1.5 × ULN； AST, ALT and alkaline phosphatase (ALP) ≤ 2.5 times the upper limit of normal value (ULN);

   Adequate renal function: serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min (calculated using Cockcroft Gault formula);
9. Sufficient coagulation function (without anticoagulation treatment): International normalized ratio (INR) ≤ 1.5;

Exclusion Criteria:

1. Have a history of hypersensitivity or intolerance to any drug used in the study;
2. Plan to receive any other anti-tumor treatment during the study period;
3. Patients who have received the second generation of androgen receptor (AR) inhibitors in the past, such as apantamide, enzalutamide, darotamide (ODM-201) or other AR inhibitors, CYP17 enzyme inhibitors, such as abietron acetate or oral ketoconazole, chemotherapy or immunotherapy, as well as adjuvant or new adjuvant therapy, should also be excluded;
4. Four weeks before the start of the study, he received plant drugs (such as saw palmetto) that have the effect of anti prostate cancer or reducing PSA level;
5. Have a history of epileptic seizures, a history of medication that can reduce the threshold of epileptic seizures, or a disease that can induce epileptic seizures within 12 months before the start of the study and treatment (including a history of transient ischemic attacks, cerebral apoplexy, brain trauma and disturbance of consciousness requiring hospitalization);
6. There were active heart diseases within 6 months before the start of study treatment, including severe/unstable angina, myocardial infarction, congestive heart failure [NYHA III or IV], or arrhythmias requiring drug treatment;
7. There is inability to swallow, chronic diarrhea, intestinal obstruction or other factors affecting drug administration and absorption;
8. Have a history of immunodeficiency (including HIV test positive, other acquired and congenital immunodeficiency diseases) or organ transplantation;
9. Known brain metastasis;
10. Malignant tumors other than prostate cancer in the past 5 years or at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
11. Those who are receiving any other experimental drugs or experimental medical devices;
12. Poor compliance, difficult to cooperate with treatment and follow-up;
13. The investigator believes that the patient has concomitant diseases (such as poorly controlled hypertension, serious diabetes, neurological or mental diseases, etc.) that seriously endanger the patient's safety, may confuse the research results, or affect the patient to complete the study, or any other situation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
3-year radiographic progression free survival (rPFS) rate | 3 years
  RPFS is defined as the time from the start of study treatment to the occurrence of imaging progress or death due to any reason, whichever occurs first.（%）

SECONDARY OUTCOMES:
Time to CRPC | 36 months
  Time to CRPC（months）
To PSA progress time; | 36 months
  Time to PSA progress（months）
Asymptomatic skeletal event (SSE) survival; | 36 months
  Asymptomatic skeletal event (SSE) survival.（%）

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No